CLINICAL TRIAL: NCT02419404
Title: Response of Pulse Pressure Variation in PA Catheter Tracing to IV Fluid Bolus in the ICU
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Robert Thiele, MD, Assistant Professor, Anesthesiology, University of Virginia
Other Study IDs: 16712
Record Dates: First submitted 2013-05-01; First posted 2015-04-17 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients having cardiac surgery: Patients having cardiac surgery who have a pulmonary artery catheter will be eligible for inclusion in this study

SUMMARY:
The investigators hypothesize that analysis of blood pressure will allow doctors to predict whether or not blood flow from the heart (cardiac output) increases after intravenous fluids are given.

DETAILED DESCRIPTION:
Total to expected enrollment: 70

ELIGIBILITY:
Inclusion Criteria:

* TCV-PO post-operative patients with PA catheters
* Must be 18 years of age and older

Exclusion Criteria:

* History of Pulmonary Hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having cardiac surgery who have a pulmonary artery catheter
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output | First five hours after surgery
  Change in cardiac output after intravenous fluids are given

CONTACTS AND LOCATIONS:
Overall Officials: ROBERT H THIELE, M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No